CLINICAL TRIAL: NCT00909922
Title: Musculoskeletal Measurements in Transfemoral Amputees
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Robert S. Gailey, PhD, PT, Miami VA Healtcare System
Other Study IDs: 3019.02
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Lower Limb Loss
Keywords: Amputation; Amputees; Artificial Limbs; Leg Length Inequality; Lower Extremity; Pelvis; Posture; Prostheses; Range of Motion; Trunk Muscles
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lower Limb Amputees: Unilateral Above knee amputees

SUMMARY:
The aim of this study was to identify posture asymmetries in transfemoral amputees utilizing clinical evaluation measures. The purposes of this investigation were: 1) to measure the limb length indirectly to determine the proportion of participants with LLD and to quantify the mean amount of discrepancy. The investigators hypothesized that a majority of transfemoral amputees would present with a short prosthetic limb. 2) To measure pelvic tilt to determine if transfemoral amputees undergo musculoskeletal adaptations similar to those reported in the literature. The investigators hypothesized that transfemoral amputees would present with a greater degree of anterior pelvic tilt and pelvic innominate asymmetry than what has been previously reported. 3) To assess restriction in lateral trunk flexion and hip extension to determine if asymmetry was present and if it was related to the increase in anterior pelvic tilt. The investigators hypothesized that restrictions would be found in the lateral trunk flexors and hip flexors on the amputated side contributing to posture asymmetry at the pelvis. 4) To determine if musculoskeletal adaptations at the pelvis were affected by prosthetic limb length, lateral trunk flexion and hip extension restrictions, and residual limb length. The investigators hypothesized that the previously reported posture asymmetries would contribute to musculoskeletal adaptations at the pelvis and trunk. Results of the present study will provide a reference for clinicians when using clinical evaluation measures to determine the presence of posture asymmetries in transfemoral amputees. If posture asymmetries are detected, clinicians need to determine musculoskeletal structures at fault and offer treatment solutions to prevent secondary impairments.

ELIGIBILITY:
Inclusion Criteria:

Healthy Individuals with:

1. Unilateral transfemoral or knee disarticulation amputations between the ages 18 to 80.
2. History of at least one episode of low back pain in the past.
3. Ambulate independently of an assisted device or those who require the use of a cane or crutches for walking on level grounds.
4. Comfortably fitted with prosthesis for a period of at least 6 months.
5. More than 12 months post-amputation.

Exclusion Criteria:

Individuals with:

1. Amputation on the contralateral limb.
2. Open wound on non-amputated side.
3. Neurological disorders such as Parkinson's disease or stroke that affect their ability to ambulate.
4. Who require a walker or wheelchair for locomotion on level ground.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unilateral Transfemoral and Knee Disarticulation Amputees
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Limb Length Discrepancy | Time of Observation
Standing Pelvic Tilt | Time of Observation
Lateral Trunk Flexion | Time of Observation
Hip Extension Range of Motion | Time of observation

SECONDARY OUTCOMES:
Residual Limb Length | Time of Observation

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Veterans Affairs Healthcare System, Miami, Florida, United States